CLINICAL TRIAL: NCT05820217
Title: External Validation of the Clinical Pre-hospital "Red- Flag" Alert for Activation of Intra-hospital Hemorrhage Control Response in Blunt Trauma. A Prospective Multicentric Study
Brief Title: External Validation of the Clinical Pre-hospital "Red- Flag" Alert for Activation of Intra-hospital Hemorrhage Control Response in Blunt Trauma.
Acronym: RED-FLAG 2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Rennes University Hospital (Other); University Hospital, Tours (Other); Hospital, Laval, France (Unknown); Hospital, Le Mans, France (Unknown); Hospital, Chambery, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RED-FLAG 2
Record Dates: First submitted 2023-03-24; First posted 2023-04-19 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Trauma Injury
Keywords: Injury; Severe haemorrhage; Severe trauma
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
External validation of the clinical pre-hospital "Red- Flag" alert for activation of intra-hospital hemorrhage control response in blunt trauma.

DETAILED DESCRIPTION:
Severe trauma, with a variety of causes, is responsible for more than 9% of the world's population and is the leading cause of preventable mortality among 15-35 year olds. Massive hemorrhage remains the second leading cause of early mortality in those traumatized after head trauma, accounting for about 40% of deaths. In 71% of cases this mortality is pre-hospital without access to rapid medicalization. Intra-hospital mortality is also important.

The main factors explaining this mortality in patients with severe bleeding are delays in recognition and management. The effectiveness of the "trauma systems" and the management channels for severe traumatized injuries are thus generally assessed by the intra-hospital mortality rate. Optimal and early management is therefore essential from the pre-hospital phase.

The treatment of traumatic hemorrhagic shock requires means of local hemostasis, medication management and can go as far as the establishment of massive transfusion protocols (PTM). This type of PTM is activated in about 8% of cases. While it is little practiced in pre-hospital and still debated today, its early hospital establishment is essential.

Rym Hamada et al. highlighted a predictive score "RED-FLAG" of severe hemorrhage in severe traumatized patients requiring the immediate implementation of rapid hemorrhage control (activation of PTM, hemostasis surgery, etc.).

This score is based on 5 clinico-biological items. A score of 2 or more is predictive of an immediate intra-hospital action of hemostasis. In France, several networks are organized around centers 15 and hospitals specialized in the management of severe traumatized, from alert to definitive treatment, in accordance with the international recommendations in force.

The objective of this study is to perform external and prospective validation, within a new cohort, of the "RED-FLAGS" score. For this, we are conducting a multicenter and prospective study

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (More than 18 yo)
* Regulated by the medical regulation centers (SAMU - centres 15) of the hospitals of Angers (SAMU 49), Rennes (SAMU 35), Le Mans (SAMU 72), Tours (SAMU 37), Laval (SAMU 53) and Chambéry (SAMU 73)
* Patients with severe trauma classified as A or B
* And benefiting respectively from hospital support in trauma centers
* Not subject to limitation of active therapeutics
* Member or beneficiary of a social security scheme

Exclusion criteria:

* Patients with Not Considered Severe Trauma (Not A, B or C) after pre-hospital medical assessment
* Patient objecting to participating in research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In France, the pre-hospital response system is organised. Any traumatized patient or witness of a trauma has the opportunity to request health assistance by calling the "15 emergency number". Under medical regulation, the emergency physician will hire pre-hospital road and/or helicopter medical means in order to medically and quickly take care of these patients.
  The collections of information will then be made by 6 centers
  This population of severely traumatized patients supported by medicalized Mobile Emergency and Resuscitation Facilities (SMUR) will be our study population. A systematic collection of information from these patients will be collected prospectively using a SMUR sheet.
Sampling Method: Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2023-05-10 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Specific intra-hospital severe haemorrhage response | 24 hours
  The main evaluation criterion is defined, as in the initial study by Hamada et al., by the presence of intrahospital criteria for severe hemorrhage justifying an immediate intrahospital action of hemostasis, defined by:
  * Red Blood Cell Concentrate transfusion required upon arrival at trauma center
  * Transfusion of at least 4 CGR within the first 6 hours of hospital management
  * Lactacidemy 5 mmol/L at first blood collection
  * Need for hemostasis surgery or radiology interventional prior to completion of a pan-body CT lesion assessment
  * Death from hemorrhagic shock within first 24 hours admission
  The ability of the RED-FLAG score to detect patients with severe hospital bleeding requiring immediate hemostasis action (as defined above) will be assessed by determining the area under the curve and its 95% CI of the ROC curve of this score.

SECONDARY OUTCOMES:
Comparison of the two RED-FLAG and BATT scores | 24 hours
  We will compare the two BATT score and the RED-FLAG scores results and their possible correlation between. We will use the Pearson linear coefficient to make the comparison.
  The BATT (Bleeding Audit for Trauma & Triage) score is a score with a minimum of 0 and a maximum of 27 points. Its identifies trauma patient at risk of significant haemorrhage. A score of 2 or more would be an appropriate threshold for pre-hospital tranexamic acid treatment.
  The RED-FLAG score is a score with a minimum of 0 and a maximum of 5 points. A score greater than or equal to 2 points identifies severe blunt trauma patients during the pre-hospital care phase and activating a specific immediate intra-hospital haemorrhage control response prior to arrival.

REFERENCES:
- [Result] Davis KA, Fabian TC, Cioffi WG. The Toll of Death and Disability From Traumatic Injury in the United States-The "Neglected Disease" of Modern Society, Still Neglected After 50 Years. JAMA Surg. 2017 Mar 1;152(3):221-222. doi: 10.1001/jamasurg.2016.4625. No abstract available. PMID 28030708
- [Result] Krug EG, Sharma GK, Lozano R. The global burden of injuries. Am J Public Health. 2000 Apr;90(4):523-6. doi: 10.2105/ajph.90.4.523. PMID 10754963
- [Result] Sauaia A, Moore FA, Moore EE, Moser KS, Brennan R, Read RA, Pons PT. Epidemiology of trauma deaths: a reassessment. J Trauma. 1995 Feb;38(2):185-93. doi: 10.1097/00005373-199502000-00006. PMID 7869433
- [Result] Beck B, Smith K, Mercier E, Gabbe B, Bassed R, Mitra B, Teague W, Siedenburg J, McLellan S, Cameron P. Differences in the epidemiology of out-of-hospital and in-hospital trauma deaths. PLoS One. 2019 Jun 4;14(6):e0217158. doi: 10.1371/journal.pone.0217158. eCollection 2019. PMID 31163036
- [Result] Baker CC, Oppenheimer L, Stephens B, Lewis FR, Trunkey DD. Epidemiology of trauma deaths. Am J Surg. 1980 Jul;140(1):144-50. doi: 10.1016/0002-9610(80)90431-6. PMID 7396078
- [Result] Shackford SR, Mackersie RC, Holbrook TL, Davis JW, Hollingsworth-Fridlund P, Hoyt DB, Wolf PL. The epidemiology of traumatic death. A population-based analysis. Arch Surg. 1993 May;128(5):571-5. doi: 10.1001/archsurg.1993.01420170107016. PMID 8489391
- [Result] Teixeira PG, Inaba K, Hadjizacharia P, Brown C, Salim A, Rhee P, Browder T, Noguchi TT, Demetriades D. Preventable or potentially preventable mortality at a mature trauma center. J Trauma. 2007 Dec;63(6):1338-46; discussion 1346-7. doi: 10.1097/TA.0b013e31815078ae. PMID 18212658
- [Result] Moore L, Stelfox HT, Evans D, Hameed SM, Yanchar NL, Simons R, Kortbeek J, Bourgeois G, Clement J, Turgeon AF, Lauzier F. Trends in Injury Outcomes Across Canadian Trauma Systems. JAMA Surg. 2017 Feb 1;152(2):168-174. doi: 10.1001/jamasurg.2016.4212. PMID 27829100
- [Result] Cameron PA, Gabbe BJ, Cooper DJ, Walker T, Judson R, McNeil J. A statewide system of trauma care in Victoria: effect on patient survival. Med J Aust. 2008 Nov 17;189(10):546-50. doi: 10.5694/j.1326-5377.2008.tb02176.x. PMID 19012550
- [Result] Abe T, Komori A, Shiraishi A, Sugiyama T, Iriyama H, Kainoh T, Saitoh D. Trauma complications and in-hospital mortality: failure-to-rescue. Crit Care. 2020 May 15;24(1):223. doi: 10.1186/s13054-020-02951-1. PMID 32414401
- [Result] Shackelford SA, Del Junco DJ, Powell-Dunford N, Mazuchowski EL, Howard JT, Kotwal RS, Gurney J, Butler FK Jr, Gross K, Stockinger ZT. Association of Prehospital Blood Product Transfusion During Medical Evacuation of Combat Casualties in Afghanistan With Acute and 30-Day Survival. JAMA. 2017 Oct 24;318(16):1581-1591. doi: 10.1001/jama.2017.15097. PMID 29067429
- [Result] Hamada SR, Rosa A, Gauss T, Desclefs JP, Raux M, Harrois A, Follin A, Cook F, Boutonnet M; Traumabase(R) Group; Attias A, Ausset S, Boutonnet M, Dhonneur G, Duranteau J, Langeron O, Paugam-Burtz C, Pirracchio R, de St Maurice G, Vigue B, Rouquette A, Duranteau J. Development and validation of a pre-hospital "Red Flag" alert for activation of intra-hospital haemorrhage control response in blunt trauma. Crit Care. 2018 May 5;22(1):113. doi: 10.1186/s13054-018-2026-9. PMID 29728151
- [Result] Ageron FX, Coats TJ, Darioli V, Roberts I. Validation of the BATT score for prehospital risk stratification of traumatic haemorrhagic death: usefulness for tranexamic acid treatment criteria. Scand J Trauma Resusc Emerg Med. 2021 Jan 6;29(1):6. doi: 10.1186/s13049-020-00827-5. PMID 33407716